CLINICAL TRIAL: NCT01517542
Title: Evaluation on the Effectiveness of Nutritional Counseling on an Adapted DASH Diet in Patients After Stroke: a Randomized Clinical Trial
Brief Title: Evaluation of Effectiveness of Nutritional Counseling in Patients After Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low availability of professionals to recruit the participants
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, SHEILA CRISTINA OURIQUES MARTINS, Principal Investigator, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-0014
Record Dates: First submitted 2011-11-22; First posted 2012-01-25 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Cardiovascular Diseases
Keywords: diet; DASH; Stroke; Nutritional counseling
MeSH Terms: conditions — Stroke; Cardiovascular Diseases | interventions — Nutrition Assessment; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional counseling (Experimental): It was composed by patients who received specific written orientation to follow the DASH diet recommendations. Calories were calculated with the goal of maintaining body weight and divided into 3 main meals and two to three snacks.
  Interventions: Other: Nutritional Counseling
- Usual diet (No Intervention): It was composed by patients who were stimulated to follow the general orientations of the neurologist or keep their food intake habits

INTERVENTIONS:
Other: Nutritional Counseling — 2 groups: 1 with nutritional counseling and other with usual diet without nutritional counseling
  Other Names: adherence; nutrition
  Arms: Nutritional counseling

SUMMARY:
Stroke is the leading cause of disability worldwide and the leading cause of death in Brazil. It is estimated that about 18 million people will have a stroke in 2015 and approximately one third of these resulting in death. The factors most important modifiable risk for stroke include high blood pressure (hypertension), diabetes, smoking, dyslipidemia, sedentary lifestyle and obesity. Acting on these risk factors can be reduced by 88% the risk of another stroke. Healthy eating is among the changes in lifestyle that are recommended for prevention and treatment of one of the main risk factors for stroke. Studies show that the adoption of the DASH diet can significantly reduce blood pressure and the result is even more significant in hypertensive patients, making this diet a new alternative in the prevention and treatment of hypertension and consequently stroke. Compliance therapy is a determining factor for success in the treatment of chronic diseases. Adherence to long-term treatment in developed countries is around 50% and in developing countries the rates are even lower. The aim of this study is to evaluate the effectiveness of nutritional counseling in an adapted DASH style diet on body weight, glycemic control, blood pressure values and improved lipid profile compared to the usual diet without nutritional counseling in patients with stroke within the last 3 months. The hypothesis is that nutritional counseling with an adapted DASH style diet reduces cardiovascular risk factors compared with the usual diet without nutritional counseling in patients with stroke within 3 months. The stroke patients will be selected in the hospitalization or in the outpatient clinic of Hospital de Clínicas de Porto Alegre in a period up to 3 months after ischemic stroke. The patients will be randomized to one of the 2 groups. In the first visit they will be submitted to a social class and international physical activity questionnaire and they will be submitted to a food frequency questionnaire, measures of weight, height, waist circumference, hip and neck, blood pressure and cholesterol and glucose measurements at the baseline, 30 days and 3, 6, 9 and 12 months. The main endpoints will be the change in the body weight, blood glucose, blood pressure values and lipid profile.

DETAILED DESCRIPTION:
The study will be followed by a evaluation of other endpoints: new stroke, myocardial infarction or cardiovascular death.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic Stroke up to 3 months
* Modified Rankin Score < 4

Exclusion Criteria:

* Aphasia
* Enteral diet
* Unavailability to follow up the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline arterial blood pressure and 6 months | 30 days and 3, 6, 9 and 12 months
  The patients will be randomized to one of the 2 groups (with nutritional counseling and no intervention - habitual diet). The main endpoint will be the change in the blood pressure values and adherence to treatment measured in 30 days and 3, 6, 9 and 12 months.

SECONDARY OUTCOMES:
Change in lipids from baseline | 30 days, 3, 6, 9 and 12 months
  The patients will be randomized to one of the 2 groups (with nutritional counseling and no intervention - habitual diet). The secundary endpoint will be the change in the lipid profile and adherence to treatment measured in 30 days and 3, 6, 9 and 12 months.
Change in the body weight | 30 days and 3, 6, 9 and 12 months
  The patients will be randomized to one of the 2 groups (with nutritional counseling and no intervention - habitual diet). The secundary endpoint will be the change in the body weight measured in 30 days and 3, 6, 9 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila CO Martins, PI, Principal Investigator — Hospital de Clínicas de Porto Alegre; Vanessa A Piper, SI, Study Director — Hospital de Clínicas de Porto Alegre; Márcia LF Chaves, SI, Study Chair — Hospital de Clínicas de Porto Alegre